CLINICAL TRIAL: NCT04278937
Title: Antenatal Azithromycin to Prevent Preterm Birth in Pregnant Women With Vaginal Cerclage. A Randomized Controlled Trial
Brief Title: Antenatal Azithromycin to Prevent Preterm Birth in Pregnant Women With Vaginal Cerclage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Lecturer, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU 1304/2019
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Preterm Birth
Keywords: cerclage; azithromycin
MeSH Terms: conditions — Premature Birth | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin group (Active Comparator): women will receive 500mg Azithromycin (Zithrokan®, Hikma, Egypt) one tablet orally twice daily for three days in 3 courses at 14 weeks, 24 weeks and 32 weeks in addition to routine usual antenatal care.
  Interventions: Drug: Azithromycin Tablets
- Control group (No Intervention): women will receive routine antenatal care without antibiotic prophylaxis after cerclage.

INTERVENTIONS:
Drug: Azithromycin Tablets — one tablet orally twice daily for three days in 3 courses at 14 weeks, 24 weeks and 32 weeks
  Other Names: Zithrokan®
  Arms: Azithromycin group

SUMMARY:
In women with indicated vaginal cerclage, this study aims to assess the efficacy of antenatal prophylactic Azithromycin in preventing preterm labor.

DETAILED DESCRIPTION:
Study procedures and interventions:

1. After approval of study protocol, pregnant women who underwent vaginal cerclage at Ain Shams University Maternity Hospital will be enrolled into the study according to inclusion and exclusion criteria.
2. Eligible patients will be randomized using a computer-generated sequence 1:1 either to the Azithromycin group or to non-Azithromycin group.

Randomization: Will be done using computer generated randomization sheet using MedCalc© version 13.

Allocation and Concealment: Will be done by use of sealed opaque envelopes that will be given to a third party (nurse) who will assign the women to study arms. Each woman will be invited to pull out an envelope. According to the number inside her envelope, women will be allocated to either group 1 or group 2 according to a computer- generated random list.

3. Intervention:

1. st group (Azithromycin group): 25 women will receive 500mg Azithromycin (Zithrokan®, Hikma, Egypt) one tablet orally twice daily for three days in 3 courses at 14wk, 24wk and 32wk in addition to routine usual antenatal care.
2. nd group (non-Azithromycin group): 25 women will receive routine antenatal care without antibiotic prophylaxis after cerclage.

4. Follow up: Through antenatal care at 4 weeks interval till 28 weeks gestational age then at 2 weeks interval till delivery.

History: Routine ANC history with special comment on history of infection as (pain, bleeding, offensive discharge).

Examination: Routine ANC examination with special comment on signs of infection (fever, tachycardia).

Investigation: As scheduled routine labs (CBC, Urine analysis, etc) and ultrasound.

5. Data collection and recording case record form: The data will be collected in a case record form (age, parity, body mass index (BMI), mode of the delivery, previous adverse perinatal outcome, gestational age at time of delivery, birth weight, NICU admission, still birth, miscarriage, antepartum hemorrhage, hospital stay, postpartum pyrexia, ICU admission, need for blood transfusion.

To decrease risk of bias, the observer collecting the data will be blinded as regards whether they are azithromycin group or non-azithromycin group.

Statistical analysis:

The collected data will be revised, coded, tabulated and introduced to a PC using Statistical package for Social Science (SPSS 20.0.1 for windows; SPSS Inc, Chicago, IL, 2001). Quantitative variables are expressed as mean and SD, or Median and Interquartile range (IQR) according to distribution of data. Qualitative variables are expressed as frequencies and percentages. Student t test and Mann Whitney Test will be used to compare a continuous variable between two study groups. Chi square test will be used to examine the relationship between Categorical variables. A P-value< 0.05 was considered statistically significant.

Ethical and Safety Consideration:

This study will be done after approval of the ethical committee of the department of obstetrics and gynecology, faculty of medicine, Ain Shams University. Informed consent will be taken from all participants before recruitment in the study, and after explaining the purpose and procedures of the study. The investigator will obtain the written, signed informed consent of each subject prior to performing any study specific procedures on the subject. The investigator will retain the original signed informed consent form. All data will be collected confidentially. Women with vaginal cerclage will be counseled about the side effects associated with cerclage and Azithromycin. The study will be based on the investigator self-funding.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age (14-34 weeks).
2. Pregnant women who underwent vaginal cerclage (either history- based or ultrasound based vaginal cerclage)

History based cerclage:

* History of one or more second-trimester pregnancy losses related to painless cervical dilatation and in absence of labor or abruptio placentae; OR
* Prior cerclage due to painless cervical dilation in the second trimester

Ultrasound based cerclage:

Current singleton pregnancy, prior spontaneous preterm birth at less than 34 weeks of gestation, and short cervical length (less than 25 mm) before 24 weeks of gestation

Exclusion Criteria:

1. Multiple pregnancy.
2. Current or past history of medical diseases (Diabetes Milletus, Hypertension, Systemic Lupus Erythematosus, Cardiac diseases, etc ).
3. Adverse perinatal outcome due to abdominal trauma.
4. Structural fetal anomalies detected during anomaly scan.
5. Allergy to Azithromycin

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Gestational age at time of delivery | At time of delivery
  the gestational age measured in weeks

SECONDARY OUTCOMES:
Birth weight | At time of delivery
  the weight of the baby measured in grams
Neonatal complications | At time of delivery and in the first postpartum week
  complications occurring in the neonate (still birth / neonatal intensive care unit admission).
Maternal complications | At time of delivery and in the first postpartum week
  complications occurring in the mother (antepartum hemorrhage, postpartum pyrexia >38 Celsius, need for blood transfusion, hospital stay, ICU admission).

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Ashoush, MD, Study Director — Professor; Hassan A Bayoumy, MD, Study Chair — Professor
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Ahmed RHM, Bayoumy HA, Ashoush SA, Gabr WKL. Antenatal azithromycin to prevent preterm birth in pregnant women with vaginal cerclage: A randomized clinical trial. Turk J Obstet Gynecol. 2023 Mar 10;20(1):1-7. doi: 10.4274/tjod.galenos.2023.47715. PMID 36907997